CLINICAL TRIAL: NCT02207491
Title: A Double-masked, Randomized, Multi-center, Active-controlled, Parallel, 3-month Study Assessing the Safety and Ocular Hypotensive Efficacy of AR-13324 Ophthalmic Solution, 0.02% Compared to Timolol Maleate Ophthalmic Solution, 0.5% in Patients With Elevated Intraocular Pressure
Brief Title: Double-masked Study of AR-13324 Ophthalmic Solution in Patients With Glaucoma or Ocular Hypertension
Acronym: Rocket-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-13324-CS301
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-01

CONDITIONS: Ocular Hypertension; Open-angle Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Glaucoma | interventions — BID protein, human; netarsudil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AR-13324 Ophthalmic Solution 0.02% & Placebo (Experimental): 1 drop AR-13324 in the evening (PM) & 1 drop placebo in the morning (AM) in both eyes (OU)
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.02%; Other: Placebo
- Timolol maleate Ophthalmic Solution 0.5% BID (Active Comparator): 1 drop Timolol maleate twice daily (BID) in the morning (AM) & evening (PM) in both eyes (OU)
  Interventions: Drug: Timolol maleate Ophthalmic Solution 0.5% BID

INTERVENTIONS:
Drug: Timolol maleate Ophthalmic Solution 0.5% BID — 1 drop BID, AM/PM, OU
  Arms: Timolol maleate Ophthalmic Solution 0.5% BID
Drug: AR-13324 Ophthalmic Solution 0.02% — 1 drop once daily (QD), PM, OU
  Other Names: Netarsudil
  Arms: AR-13324 Ophthalmic Solution 0.02% & Placebo
Other: Placebo — 1 drop QD, AM, OU
  Arms: AR-13324 Ophthalmic Solution 0.02% & Placebo

SUMMARY:
To evaluate the ocular hypotensive efficacy and ocular and systemic safety of AR-13324 Ophthalmic Solution, 0.02% compared to the active comparator Timolol maleate Ophthalmic Solution, 0.5%

ELIGIBILITY:
Subject Inclusion criteria:

1. 0-2 years of age and 18 years or greater.
2. Diagnosis of open angle glaucoma or ocular hypertension
3. Unmedicated (post-washout) IOP (Intraocular Pressure) >20 mm Hg and < 27 mm Hg in the study eye at 2 qualification visits.
4. Corrected visual acuity in each eye equivalent to 20/200.
5. Able and willing to give signed informed consent (parent or guardian consent for pediatric patient) and follow study instructions.

Subject exclusion criteria

Ophthalmic:

1. Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure, or narrow angles. Note: Previous laser peripheral iridotomy is NOT acceptable.
2. Intraocular pressure ≥27 mm Hg (unmedicated) in both eyes (individuals who are excluded for this criterion are not allowed to attempt requalification), or use of more than two ocular hypotensive medications within 30 days of screening. Note: fixed dose combinations count as two medications.
3. Known hypersensitivity to any component of the formulations to be used (benzalkonium chloride, etc.), to topical anesthetics or beta adrenoceptor antagonists.
4. Previous glaucoma intraocular surgery or glaucoma laser procedures in either eye
5. Refractive surgery in either eye.
6. Ocular trauma in either eye within the six months prior to screening, or ocular surgery or non-refractive laser treatment within the three months prior to screening.
7. Recent or current evidence of ocular infection or inflammation in either eye. Current evidence of clinically significant blepharitis, conjunctivitis, or a history of herpes simplex or zoster keratitis at screening in either eye.
8. Ocular medication in either eye of any kind within 30 days of screening.
9. Clinically significant ocular disease in either eye (e.g., corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe.
10. Central corneal thickness in either eye greater than 600 µm at screening.
11. Any abnormality in either eye preventing reliable applanation tonometry of either eye.

    Systemic:
12. Clinically relevant abnormalities (as determined by the investigator) in laboratory tests at screening which may impact the study.
13. Known hypersensitivity or contraindication to beta-adrenoceptor antagonists (e.g., chronic obstructive pulmonary disease or bronchial asthma; abnormally low blood pressure or heart rate; second or third degree heart block or congestive heart failure; severe diabetes).
14. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study.
15. Participation in any investigational study within 30 days prior to screening.
16. Changes of systemic medication that could have an effect on intraocular pressure within 30 days prior to screening, or anticipated during the study.
17. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the screening examination and must not intend to become pregnant during the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Heah, MD, Study Director — Aerie Pharmaceuticals, Inc.
Locations (1):
- Aerie Pharmaceuticals, Bedminster, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 35 clinical trial sites starting in June of 2014. The first participant was enrolled in July of 2014 and the last participant was enrolled in December of 2014.
Pre-assignment Details: Prior to enrollment, adult participants were to have a Screening Visit and 2 Qualification Visits to allow for washout of ocular hypotensive medication if needed.
  The Randomized Population includes all subjects who were randomized to treatment. Baseline variables and demographic characteristics were summarized for this population.
Groups:
- Timolol Maleate Ophthalmic Solution 0.5% BID: 1 drop Timolol maleate twice daily (BID) in the morning (AM) and evening (PM) in both eyes (OU)
Period: Overall Study
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID
Started | 202 | 209
Completed | 171 | 196
Not Completed | 31 | 13
Not completed — Adverse Event | 20 | 4
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Non-compliant | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 3 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 3 | 5

BASELINE CHARACTERISTICS:
Population: Randomized Population
Groups:
- Total: Total of all reporting groups
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID | Total
Number analyzed (Participants) | 202 | 209 | 411
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (11.65) | 64.2 (11.34) | 65.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 136 | 250
  Male | 88 | 73 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 28 | 55
  Not Hispanic or Latino | 175 | 181 | 356
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 51 | 94
  White | 157 | 153 | 310
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: The primary efficacy outcome is mean IOP
Time Frame: 3 months
Population: Per-Protocol (PP) Population. The PP population includes subjects who did not have major protocol violations likely to seriously affect the primary outcome of the study. The PP population summarizes subjects as treated for purpose of analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID
Number analyzed (Participants) | 182 | 188
mmHg
  Day 1, 0800 hours | 23.42 (1.756) | 23.37 (1.658)
  Day 1, 1000 hours | 22.28 (2.128) | 21.92 (2.053)
  Day 1, 1600 hours | 21.78 (2.385) | 21.45 (2.365)
  Day 15, 0800 hours: number analyzed (Participants) | 177 | 187
  Day 15, 0800 hours | 18.68 (3.342) | 18.33 (2.566)
  Day 15, 1000 hours: number analyzed (Participants) | 176 | 186
  Day 15, 1000 hours | 17.29 (3.303) | 17.55 (2.570)
  Day 15, 1600 hours: number analyzed (Participants) | 176 | 186
  Day 15, 1600 hours | 17.24 (3.294) | 17.70 (2.661)
  Day 43, 0800 hours: number analyzed (Participants) | 170 | 184
  Day 43, 0800 hours | 19.35 (3.629) | 18.24 (2.924)
  Day 43, 1000 hours: number analyzed (Participants) | 170 | 184
  Day 43, 1000 hours | 18.14 (3.502) | 17.44 (2.725)
  Day 43, 1600 hours: number analyzed (Participants) | 170 | 183
  Day 43, 1600 hours | 17.86 (3.580) | 17.71 (2.820)
  Day 90 (month 3), 0800 hours: number analyzed (Participants) | 157 | 181
  Day 90 (month 3), 0800 hours | 19.81 (3.647) | 18.47 (2.711)
  Day 90 (month 3), 1000 hours: number analyzed (Participants) | 158 | 181
  Day 90 (month 3), 1000 hours | 18.92 (3.702) | 17.96 (2.674)
  Day 90 (month 3), 1600 hours: number analyzed (Participants) | 158 | 181
  Day 90 (month 3), 1600 hours | 18.48 (3.595) | 17.74 (2.546)
Statistical Analysis 1: Comparison: AR-13324 Ophthalmic Solution 0.02% & Placebo vs Timolol Maleate Ophthalmic Solution 0.5% BID; Assuming zero difference between AR-13324 and timolol, a 2-tailed alpha of 0.05 at each of 9 time points, a common SD of 3.0 mmHg, and a correlation between time points of 0.60 or less, 170 PP subjects per arm were necessary to have 90% power to show clinical noninferiority of AR-13324 to timolol in mean IOP; Test type: Non-Inferiority — Clinical noninferiority was to be concluded if the upper limit of the 95% CIs around the difference (AR-13324 - timolol) was within 1.5 mmHg at all time points and was within 1.0 mmHg at a majority of the time points; p < 0.0001, ANCOVA — Calculated p-value; Statistical analysis applies at all 3 timepoints on Day 15, Day 43, and Day 90

2. Secondary Outcome: Extent of Exposure
Description: Exposure to study medication in days for all treatment groups.
Time Frame: 3 months
Population: Safety Population: all randomized subjects who received at least 1 dose of study medication. The safety population summarizes subjects as treated for purpose of analysis. Three (3) subjects received incorrect study medication from that to which they were randomized, shown in the Participant Flow.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID
Number analyzed (Participants) | 203 | 208
days | 82.8 (21.44) | 87.4 (15.53)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the course of the 90-day treatment period.
Description: The Safety Population included all randomized subjects who received at least 1 dose of study medication and was used to summarize safety variables. Three (3) subjects received incorrect study medication from that to which they were randomized, shown in the Participant Flow.
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | Timolol Maleate Ophthalmic Solution 0.5% BID
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/208
Serious Adverse Events (participants affected / at risk) | 3/203 | 4/208
Other Adverse Events (participants affected / at risk) | 145/203 | 75/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AR-13324 Ophthalmic Solution 0.02% & Placebo (N=203) | Timolol Maleate Ophthalmic Solution 0.5% BID (N=208)
Worsening of Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Left Upper Extremity Numbness (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (CVA) (Nervous system disorders) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Exacerbation of Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AR-13324 Ophthalmic Solution 0.02% & Placebo (N=203) | Timolol Maleate Ophthalmic Solution 0.5% BID (N=208)
Conjunctival hyperemia (Eye disorders) | 108 | 17
Conjunctival Haemmorrhage (Eye disorders) | 32 | 2
Cornea Verticillata (Eye disorders) | 12 | 0
Erythema of Eyelid (Eye disorders) | 12 | 0
Vision Blurred (Eye disorders) | 11 | 1
Instillation Site Pain (General disorders) | 30 | 42
Instillation Site Erythema (General disorders) | 24 | 4
Vital Dye Staining Cornea Present (Investigations) | 17 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No